CLINICAL TRIAL: NCT02764008
Title: The Comparison of Low Thoracic Paravertebral Block Versus Peritubal Infiltration in Patients Undergoing Percutaneous Nephrolithotomy
Brief Title: The Comparison of Low Thoracic Paravertebral Block Versus Peritubal Infiltration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ahmet Murat Yayik, MD, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUTF ANESTHESIA2
Record Dates: First submitted 2016-05-04; First posted 2016-05-05 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Percutaneous Nephrolithotomy
Keywords: Postoperative Analgesia; Peritubal infiltration; Ultrasound guided low thoracic paravertebral block; Percutaneous Nephrolithotomy pain
MeSH Terms: interventions — Bupivacaine; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low thoracic paravertebral block (Active Comparator): T8-T9 Ultrasound guided paravertebral block with 20 ml %0,25 bupivacaine
  Interventions: Drug: Bupivacaine; Device: Ultrasound
- Peritubal infiltration (Active Comparator): Peritubal infiltration with 20 ml %0,25 bupivacaine
  Interventions: Drug: Bupivacaine
- Control Group (No Intervention): No drug

INTERVENTIONS:
Drug: Bupivacaine — 20 ml %0,25 bupivacaine
  Arms: Low thoracic paravertebral block; Peritubal infiltration
Device: Ultrasound
  Arms: Low thoracic paravertebral block

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is a safe and effective procedure that is considered the standard treatment for large and complex renal stones. Although it has lower complication and morbidity rates than open surgery, the pain and discomfort related to a nephrostomy tube can cause distress for patients.

Managing this pain with opioids can lead to sedation, nausea, vomiting, and constipation, which defeat the purpose of this minimally invasive procedure.

Skin infiltration with bupivacaine around the nephrostomy tube is not effective. Infiltration of renal capsule has shown to facilitate painless insertion of nephrostomy tube, suggesting the role of renal capsule in pain management.

Peritubal infiltration of bupivacaine from renal capsule to the skin along the nephrostomy tract may alleviate postoperative pain. A unilateral Low thoracic paravertebral (PVB) block offers the option of providing extendable perioperative pain relief without the above side effects or the physiologic derangement associated with local anesthetics in the central neuraxial space.

The aim of this study is to determine whether ultrasound guided low thoracic paravertebral block effective post-operative analgesia as compared to peritubal infiltration analgesia in patients undergoing percutaneous nephrolithotomy.

Main outcome measures: The primary endpoint is postoperative opioid consumption. Secondary endpoints are visual analogue pain scores, opioid related side effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients undergoing percutaneous nephrolithotomy

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications
* emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | First 24 hours total opioid consumption

SECONDARY OUTCOMES:
Visual analog pain score | postoperative first hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at first hour postoperatively.
Visual analog pain score | postoperative second hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at second hour postoperatively.
Visual analog pain score | postoperative 4th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 4th hour postoperatively
Visual analog pain score | postoperative 8th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 8th hour postoperatively
Visual analog pain score | postoperative 12th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS)score of 0-10 (0= no pain and 10= worst imaginable pain) at 12th hour postoperatively.
Visual analog pain score | postoperative 24th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS)score of 0-10 (0= no pain and 10= worst imaginable pain) at 24th hour postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ahiskalioglu, Ass.Prof., Study Director — Ataturk University Anesthesiology and Reanimation
Locations (1):
- Ataturk University, Yakutiye, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kirac M, Tepeler A, Bozkurt OF, Elbir F, Ozluk C, Armagan A, Unsal A, Biri H. The efficacy of bupivacaine infiltration on the nephrostomy tract in tubeless and standard percutaneous nephrolithotomy: a prospective, randomized, multicenter study. Urology. 2013 Sep;82(3):526-31. doi: 10.1016/j.urology.2013.02.083. Epub 2013 Jul 4. PMID 23831069
- [Background] Ak K, Gursoy S, Duger C, Isbir AC, Kaygusuz K, Ozdemir Kol I, Gokce G, Mimaroglu C. Thoracic paravertebral block for postoperative pain management in percutaneous nephrolithotomy patients: a randomized controlled clinical trial. Med Princ Pract. 2013;22(3):229-33. doi: 10.1159/000345381. Epub 2012 Dec 14. PMID 23257888